CLINICAL TRIAL: NCT03937427
Title: Unified Airway Model: Comparison of the Microbiome of the Upper and Lower Airways in Chronic Rhinosinusitis and Asthma Patients
Brief Title: Unified Airway Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Andrew Thamboo, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H16-01176
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Asthma
MeSH Terms: conditions — Disease; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRS with Asthma
- CRS without Asthma

SUMMARY:
Chronic rhinosinusitis (CRS) impacts approximately 5% of Canadians. CRS patients suffer from a combination of symptoms that include facial pain, nasal obstruction, hyposmia and mucopurulence discharge. Asthma may additionally worsen quality of life and many patients suffer from both conditions. The unified airway model illustrates a link between both conditions as tissue from the middle ear to the sinus cavity to the lungs function as one unit. Despite evidence for the unified airway model in the setting of CRS and asthma, there are no studies to our knowledge that have evaluated the microbiome (the resident microbes and their genetic expressions that affect disease) of the upper and lower airways in this patient population. Determining the microbiome of the upper and lower airways in patients suffering from CRS and asthma will further support the unified airway model but more importantly, will help contribute to understanding the pathophysiology of this inflammatory process and may help guide future management.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Able to speak and understand English
* Diagnosed with chronic rhinosinusitis with or without asthma and COPD or with a sinonasal tumor
* Undergoing sinus surgery in St Paul's Hospital

Exclusion Criteria:

* Oral antibiotics in the past month prior to surgery;
* Immunocompromised;
* Prior lung transplants;
* Known sinonasal or bronchial tumors, current or previous;
* Smoking;
* Known bleeding disorders:
* Deemed unfit by the rhinologists/respirologist for bronchoscopy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will analyze and compare the upper and lower airways from 12 CRS with asthma patients and 12 CRS without asthma patients matched for age, sex and degree of sinus disease based on CT grading using Lund-Mackay staging system.14
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-01-16; Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Pathology (histological assessment) | 1 day
  Objective is to characterize the pathology (histological assessment) of 'diseased' and 'non-diseased' tissue in CRS patients undergoing sinus surgery as assessed by their pre-surgery CT scan results and stratify based on comorbid lung disease
Gene Expression Patterns | 1 day
  Objective is to compare the upper and lower airway pathology and gene expression patterns with in patients with CRS +/- asthma compare to non-CRS patients

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Thamboo, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, B.C., Canada

IPD SHARING:
Plan to Share IPD: No